

## **Questionnaire Consent Statement**

## INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

What Women Want: Real Time Results for Screening Mammography in the Era of Patient-Experience Driven Care 2020-0980

Study Chair: Dr. Megan Kalambo, MD

The goal of this research study is to learn why patients may want to receive real-time imaging results during a screening mammogram appointment at an MD Anderson breast imaging center. Real-time imaging results means you receive the results of the mammogram right away during the same clinic visit.

If you agree to take part in this research study, you will complete a confidential, online survey about receiving real-time imaging results (for example, why you did or did not choose to receive real-time results, and if you would be willing to receive real-time results if there was a fee to receive them). You will also be asked questions about your demographics (such as age, ethnicity, and education level) and if you have a family history of breast cancer.

The survey is 16 questions long and should take less than 5 minutes to complete. Your participation in this research will be complete when you submit your survey answers.

The data collected from the survey will be kept confidential. Your responses will not be linked to you. Collected data will only be shared in aggregate form (meaning it will be put together with all other responses). Although there is a risk that you may be identified from your response to the demographic questions, no attempt will be made by the research staff to identify you.

Questionnaires may contain questions that are sensitive in nature. You may refuse to answer any question that makes you feel uncomfortable. If you have concerns about completing the questionnaire, you are encouraged to contact your doctor or the study chair.

There is no cost to you for taking part in this study. There are no benefits for you in this study. Your participation is completely voluntary. You may choose not to take part in this study.

## **Consent Questionnaire Statement**

NCT04794816 Protocol 2020-0980 November 9, 2020 Page 2 of 2

You have read the description of the study, and you have decided to participate in the research project described here. You understand that you may refuse to answer any (or all) of the questions at this or any other time. If you do not want to answer a question, you can skip the question.

During the course of this study, the research team at The University of Texas MD Anderson Cancer Center (MD Anderson) will be collecting information about you that they may share with health authorities, study monitors who check the accuracy of the information, and/or individuals who put all the study information together in report form. By answering the questions, you are providing authorization for the research team to use and share your information at any time. If you do not want to authorize the use and disclosure of your information, you may choose not to answer these questions. There is no expiration date for the use of this information as stated in this authorization.

You may withdraw your authorization at any time, in writing, for any reason as long as that information can be connected to you. You can learn more about how to withdraw your authorization by calling 713-792-6477 or by contacting the study doctor, Dr. Megan Kalambo, at 713-745-4555.

Please note that by clicking on the link, completing the survey, and submitting the survey you are providing your informed consent and authorization and agree to participate in this study.

Click here to take the Survey

http://mdanderson.co1.qualtrics.com/jfe/form/SV\_5BDJ04tkiVbl9e5